CLINICAL TRIAL: NCT01111669
Title: Intravenous Tranexamic Acid and Intraoperative Visualization During Functional Endoscopic Sinus Surgery: A Double Blind Randomized Controlled Trial
Brief Title: Intravenous Tranexamic Acid and Intraoperative Visualization During Functional Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Morgan Langille, MD, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200901
Record Dates: First submitted 2009-09-15; First posted 2010-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Rhinosinusitis With Polyposis; Chronic Hyperplastic Sinusitis
Keywords: Functional Endoscopic Sinus Surgery; Tranexamic Acid
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Patients in the tranexamic acid (TA) group will receive a bolus of TA, prepared according to patient weight (15mg / kg loading dose). The patients would also receive a continuous infusion of 1mg / kg per hour or TA preparation for the duration of the operation.
  Interventions: Drug: Tranexamic Acid
- Normal Saline (Placebo Comparator): The patients receiving placebo will receive an infusion of normal saline of the same volume of IV solution as the intervention group. Patients will receive the saline infusion on call to the operating room, approximately 30 minutes before onset of the operation. The patients would also receive a continuous infusion of normal saline for the duration of the operation.
  Interventions: Drug: Normal Saline (placebo)

INTERVENTIONS:
Drug: Tranexamic Acid — The bolus of TA is prepared according to patient weight (10mg / kg loading dose). The patients receiving placebo will receive an infusion of normal saline of the same volume of IV solution. Patients will receive the TA or saline infusion on call to the operating room, approximately 30 minutes before onset of the operation. The patients would also receive a continuous infusion of 1mg / kg per hour or TA preparation or normal saline for the duration of the operation.
  Other Names: cyklokapron
  Arms: Tranexamic Acid
Drug: Normal Saline (placebo) — The patients receiving placebo will receive an infusion of normal saline of the same volume of IV solution. Patients will receive the saline infusion on call to the operating room, approximately 30 minutes before onset of the operation. The patients would also receive a continuous infusion of saline for the duration of the operation.
  Arms: Normal Saline

SUMMARY:
Functional endoscopic sinus surgery (FESS) is an effective treatment of sinus disease. FESS is carried out using cameras to view the surgical field. Bleeding during the surgery can lead to poor surgical field visualization. Poor visualization has been associated with worse surgical outcomes. Tranexamic acid is a safe and effective agent used to achieve hemostasis during operative procedures. The current study is a randomized controlled trial in patients undergoing FESS to compare the effects of tranexamic acid versus placebo and the effects on surgical field visualization and adverse events.

DETAILED DESCRIPTION:
Study Objectives: The current study will assess the effect of tranexamic acid on intraoperative bleeding and surgical outcomes during functional endoscopic sinus surgery.

Background: Tranexamic acid is an antifibrinolytic that prevents the activation of plasminogen to plasmin. Plasmin is responsible for the degradation of fibrin clots. This is the mechanism by which tranexamic acid prevents blood clot breakdown and reduces operative bleeding. Functional endoscopic sinus surgery, or FESS, is a widely used surgical technique to treat sinusitis and other diseases of the nose and nasal cavities. Bleeding during FESS can hinder surgical progress and has been associated with an increase in complications.

Methods: The current study is randomized, double-blind and placebo- controlled. Study sample size will be calculated based on a previous study of topical intranasal TA. Participants undergoing functional endoscopic sinus surgery will be recruited for the study during a preoperative outpatient clinic visit. Each participant will be randomized to a group receiving either tranexamic acid or normal saline bolus immediately prior to the operation. Inclusion criteria for the study are as follows: patients must be diagnosed with either 1. Chronic rhinosinusitis with polyposis (CRSwP) or 2. Chronic hyperplastic sinusitis. Patients must have an ASA classification of I or II and must be undergoing bilateral FESS as treatment for one of the above diagnoses. Exclusion criteria include patients with hypertension (treated or untreated), thrombotic diathesis, vascular disease, risk factors for vascular disease, colorblindness, renal failure, and those who may be pregnant. These exclusion criteria are based on the potential risks of using tranexamic acid in these patients (see safety data information section below). The exclusion criteria for hypertension will include anyone who has been diagnosed previously with hypertension or has been on anti-hypertensive medications for this diagnosis. The hypertensive patients will be excluded due to the difficulties maintaining standardized anesthesia protocol (such as mean arterial pressure) in these patients. The authors of the current study will not be testing for pregnancy. Patients will be asked the date of their last menstrual period as per the standard pre-operative questionnaire, any patients who may be pregnant would not only be excluded from the trial but would not undergo a general anesthetic for an elective procedure due to the risk of preterm labour. The diagnosis of renal failure will be determined by patient history, the current study will not require systematic lab diagnosis to calculate renal function. The study will keep a record of the surgeon(s) and residents present during surgery to evaluate potential differences during the data analysis. The study will blind both the surgeon(s) and anesthesiologist as to what each patient received. The day before a scheduled operation of a patient enrolled in the study, the pharmacy will determine if the patient is to receive TA or placebo based on the randomization table. The bolus of TA is prepared according to patient weight (15mg/kg loading dose). The patients receiving placebo will receive an infusion of normal saline of the same volume. Patients will receive the TA or saline infusion on call to the operating room, approximately 30 minutes before onset of the operation. The patients would also receive a continuous infusion of 1mg/kg per hour or TA preparation or normal saline for the duration of the operation. The current study will use a standardized anesthesia protocol using universally accepted parameters. The operation will be carried out using primarily inhalational anesthetic. End- tidal CO2 will be maintained between the target ranges of 30-35 mmHg. The head of the bed will be elevated to 15 degrees. The target range for the mean arterial pressure will be 60-70 mmHg.

Outcome Measures: The outcome measures for the current study are as follows: 1. The Wormald grading scale, this is a validated instrument used to assess intraoperative bleeding during video endoscopy sinus surgery. Dr. Wright will apply the Wormald grading scale intraoperatively. 2. Perioperative Sinus Endoscopy (POSE) scoring system, a systematic visualization evaluation of the sinuses. 3. Lund- Kennedy endoscopic reporting system, a validated staging system for sinus disease. 4. Lund- MacKay CT score, used for radiologic evaluation of sinus disease, 5. Number of sinuses and which sinuses were involved in the operative procedure. 6. Surgical time. 7. Total blood loss (monitoring of suctioned blood and monitoring of sponges and throat packs used during the operation. 8. Completeness of the surgical procedure as affected by bleeding.

ELIGIBILITY:
Inclusion Criteria:

Patients must be diagnosed with either:

1. Chronic rhinosinusitis with polyposis (CRSwP) or
2. Chronic hyperplastic sinusitis. Patients must have an ASA classification of I or II and must be undergoing bilateral FESS as treatment for one of the above diagnoses.

Exclusion Criteria:

1. Hypertension (treated or untreated)
2. Thrombotic diathesis
3. Vascular disease, risk factors for vascular disease,
4. Colorblindness
5. Renal failure
6. Pregnancy

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The Wormald grading scale, this is a validated instrument used to assess intraoperative bleeding during video endoscopy sinus surgery. | Intraoperatively (as infusion of tranexamic acid or placebo is being infused)

SECONDARY OUTCOMES:
Perioperative Sinus Endoscopy (POSE) scoring system, a systematic visualization evaluation of the sinuses | Intraoperatively
Surgical time. | Intraoperatively
Total blood loss (monitoring of suctioned blood and monitoring of sponges and throat packs used during the operation) | Intraoperatively
Completeness of the surgical procedure as affected by bleeding. | Intraoperatively
Number and types of any complications or adverse events | Peri-operative period

CONTACTS AND LOCATIONS:
Overall Officials: Erin Wright, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, McClelland B, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD001886. doi: 10.1002/14651858.CD001886.pub2. PMID 17943760
- [Background] Ho KM, Ismail H. Use of intravenous tranexamic acid to reduce allogeneic blood transfusion in total hip and knee arthroplasty: a meta-analysis. Anaesth Intensive Care. 2003 Oct;31(5):529-37. doi: 10.1177/0310057X0303100507. PMID 14601276
- [Background] Snir M, Axer-Siegel R, Buckman G, Yassur Y. Central venous stasis retinopathy following the use of tranexamic acid. Retina. 1990;10(3):181-4. PMID 2236942
- [Background] Kitamura H, Matsui I, Itoh N, Fujii T, Aizawa M, Yamamoto R, Okuno A, Okazaki Y, Fujita Y, Kuwayama Y, Imai E, Fujii M. Tranexamic acid-induced visual impairment in a hemodialysis patient. Clin Exp Nephrol. 2003 Dec;7(4):311-4. doi: 10.1007/s10157-003-0254-y. PMID 14712363
- [Background] Kavanagh GM, Sansom JE, Harrison P, Warwick JA, Peachey RD. Tranexamic acid (Cyklokapron)-induced fixed-drug eruption. Br J Dermatol. 1993 Feb;128(2):229-30. doi: 10.1111/j.1365-2133.1993.tb15161.x. No abstract available. PMID 8457462
- [Background] Carrion-Carrion C, del Pozo-Losada J, Gutierrez-Ramos R, de Lucas-Laguna R, Garcia-Diaz B, Casado-Jimenez M, Esperanza-Jimenez Caballero ME. Bullous eruption induced by tranexamic acid. Ann Pharmacother. 1994 Nov;28(11):1305-6. doi: 10.1177/106002809402801121. No abstract available. PMID 7849353